CLINICAL TRIAL: NCT04511169
Title: A Self-guided Internet-delivered Intervention for Adults With ADHD: Study Protocol for a Micro-randomized Trial Investigating the Use of Reminders
Brief Title: MyADHD-digital Training for Adults With ADHD
Acronym: MINADHD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Haukeland University Hospital (Other)
Collaborators: University of Bergen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Treatment
Other Study IDs: 90483
Record Dates: First submitted 2020-06-17; First posted 2020-08-13 (Actual); Last update posted 2021-08-25 (Actual); Status verified 2020-05

CONDITIONS: ADHD - Combined Type

STUDY DESIGN:
Who Masked: Participant
Masking Description: The assessor do not know if the participant is randomized to remainders or not
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- remainder (Experimental): The participants who are inactive for more than 48 hours after recieving new content will recieve a remainder, in the format of a text message and an email.
  Interventions: Behavioral: digital self-help
- non-remainder (No Intervention): The participants who are inactive for more than 48 hours after recieving new content will NOT recieve a remainder, in the format of a text message and an email.

INTERVENTIONS:
Behavioral: digital self-help — The digital self-help program is targeting every-day ADHD symptoms in adults with a diagnosed ADHD
  Other Names: remainders
  Arms: remainder

SUMMARY:
Background: Attention deficit hyperactivity disorder (ADHD) is a neurodevelopmental disorder characterized by symptoms of inattention and/or hyperactivity/impulsivity that are persistent across situations and time. ADHD in adulthood, with an estimated prevalence of 2 - 3 %, is associated with challenges that may have severe consequences on their daily life functioning. Still, the availability of evidence-based psychological interventions is limited. Interventions delivered over the Internet is promising, because it may increase the availability of effective psychological interventions for a larger group of adults with ADHD. However, studies show that lack of sustained adherence is a challenge in self-guided internet interventions. Digital reminders may help increase adherence and engagement in these interventions.

DETAILED DESCRIPTION:
Background: Attention deficit hyperactivity disorder (ADHD) is a neurodevelopmental disorder characterized by symptoms of inattention and/or hyperactivity/impulsivity that are persistent across situations and time. ADHD in adulthood, with an estimated prevalence of 2 - 3 %, is associated with challenges that may have severe consequences on their daily life functioning. Still, the availability of evidence-based psychological interventions is limited. Interventions delivered over the Internet is promising, because it may increase the availability of effective psychological interventions for a larger group of adults with ADHD. However, studies show that lack of sustained adherence is a challenge in self-guided internet interventions. Digital reminders may help increase adherence and engagement in these interventions.

Objectives: The overall aim of this study is to investigate adherence and effects of a self-guided Internet-delivered intervention for adults with an ADHD diagnosis. More detailed, we will examine whether the use of reminders will increase adherence and engagement in the intervention, and consequently how this affect intervention effects.

Methods: The study uses a micro-randomized design. A total of 100 participants with an ADHD diagnosis will be included. Primary measure is adherence (completed modules) and participant feedback regarding self-reported engagement. Secondary clinical outcomes: inattention and hyperactivity/impulsivity measured by two subscales from the Adult ADHD Self-Rating Scale (ASRS); quality of life measured by Adult ADHD Quality of Life Measure (AAQol); stress measured by the Perceived Stress Scale (PSS); cognitive functioning measured with the Perceived Deficit Questionnaire (PDQ-5), and self-compassion measured by the Self compassion-Scale - short form (SCS-SF). We will use quantitative statistical procedures and qualitative methods to analyze the data.

Discussion: The results from the study will contribute to the growing research on Internet-delivered interventions. The expected results may have a major impact on further development of treatment options for adults with ADHD. Moreover, investigating ways to increase adherence in online self-guided programs could be of great value when implementing such intervention into routine care.

ELIGIBILITY:
Inclusion Criteria:

* Adults with a diagnosis of ADHD
* Access to a computer, smartphone and the Internet.
* Speaks, writes and read Norwegian

Exclusion Criteria:

* Current self-reported diagnosis of severe psychiatric illness (ongoing substance abuse, suicidal ideation or psychosis).
* Ongoing psychological treatment for ADHD or other psychiatric illnesses.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2020-05-20 (Actual); Primary Completion 2021-02-20 (Actual); Study Completion 2021-03-01 (Actual)

PRIMARY OUTCOMES:
number of remainders | up to 8 weeks
  number of remainders

SECONDARY OUTCOMES:
The Adult ADHD Self-Rating Scale | up to 40 weeks
  includes all the 18 symptoms of ADHD included in the diagnostic manual (DSM-5). ASRS is a self-report scale with 18 items, and is divided into two subscales; one scale measuring problems with Inattention (9 questions), and one scale measuring problems with Hyperactivity (9 questions). 0 to 16 means unlikely to have ADHD, 17 to 23 means likely to have ADHD, and 24 to 36 means highly likely to have ADHD
Adult ADHD Quality of Life Measure | up to 40 weeks
  Each item is rated by participant s on a five-point Likert scale ranging from "Not at all/ Never" (1) to "Extremely/Very Often" (5).
The perceived stress scale | up to 40 weeks
  The Perceived Stress Scale (PSS) is a widely used psychological instrument for measuring stress. Items were designed to measure stress and how uncontrollable respondents find their lives during the last month (Cohen et al, 1983). The PSS version used in this study has 10 items with response alternatives 0 (never) to 4 (very often) and an internal reliability of a Cronbach's alpha of 0.89 (Roberti et al, 2006)
The Patient Health Questionnaire-9 | up to 40 weeks
  The Patient Health Questionnaire-9 (PHQ-9: Kroenke et al., 2001) is a self-report tool used to assess the presence and severity of depressive symptoms. Reliability and validity of the tool have indicated it has sound psychometric properties. Internal consistency of the PHQ-9 has been shown to be high
The self-compassion scale - short form | up to 40 weeks
  The scale includes 6 subscales that measure how often people respond to feelings of inadequacy or suffering with self-kindness, self-judgment, common humanity, isolation, mindfulness and over-identification. Questions are rated on a scale from 1 (almost never) to 5 (almost always).
The Perceived Deficits Questionnaire 5-item | up to 40 weeks
  brief assessment of subjective cognitive difficulties and covers problems with concentration (e.g. "trouble concentrating on things like watching a television program or reading a book?"), memory (e.g. "forget what you talked about after a telephone conversation?"), and executive functioning (e.g. "have trouble getting things organized?"). Every item is rated on a scale of 0 (Never) to 4 (Almost always) to yield a sum score of 0 to 20, with higher scores indicating greater severity of cognitive symptoms.

CONTACTS AND LOCATIONS:
Locations (1):
- Community Sample, Bergen, Norway

IPD SHARING:
Plan to Share IPD: Undecided
we will share interaction data. not decided regarding health-related data

REFERENCES:
- [Derived] Nordby ES, Guribye F, Nordgreen T, Lundervold AJ. Silver linings of ADHD: a thematic analysis of adults' positive experiences with living with ADHD. BMJ Open. 2023 Oct 3;13(10):e072052. doi: 10.1136/bmjopen-2023-072052. PMID 37788928
- [Derived] Kenter RMF, Schonning A, Inal Y. Internet-Delivered Self-help for Adults With ADHD (MyADHD): Usability Study. JMIR Form Res. 2022 Oct 21;6(10):e37137. doi: 10.2196/37137. PMID 36269662
- [Derived] Nordby ES, Gjestad R, Kenter RMF, Guribye F, Mukhiya SK, Lundervold AJ, Nordgreen T. The Effect of SMS Reminders on Adherence in a Self-Guided Internet-Delivered Intervention for Adults With ADHD. Front Digit Health. 2022 May 16;4:821031. doi: 10.3389/fdgth.2022.821031. eCollection 2022. PMID 35651537
- [Derived] Flobak E, Nordby ES, Guribye F, Kenter R, Nordgreen T, Lundervold AJ. Designing Videos With and for Adults With ADHD for an Online Intervention: Participatory Design Study and Thematic Analysis of Evaluation. JMIR Ment Health. 2021 Sep 14;8(9):e30292. doi: 10.2196/30292. PMID 34519666